CLINICAL TRIAL: NCT07321379
Title: Efficacy of Bicarbonate on the Risk of Assisted Delivery in Danish Nulliparous Women With Prolonged Labour: a Double-blinded Parallel Randomized Controlled Trial (The ProLabour Trial)
Brief Title: Efficacy of Bicarbonate on the Risk of Assisted Delivery in Nulliparous Women With Prolonged Labour
Acronym: ProLabour
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: University of Copenhagen (Other); Rigshospitalet, Denmark (Other); Aarhus University Hospital (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); University of Liverpool (Other); University of Amsterdam (Other)
Responsible Party: Principal Investigator, Nanna Maaløe, Associate Professor, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-0338
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Prolonged Labor; Labor Dystocia
Keywords: Labor; Bicarbonate; Caesarean section; Assisted birth; Oxytocin; Labor augmentation; Intrapartum
MeSH Terms: conditions — Dystocia | interventions — Sodium Bicarbonate

STUDY DESIGN:
Intervention Model Description: The Danish ProLabour Trial is a double-blinded, parallel group, randomized-controlled, superiority trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The active substance, sodium bicarbonate, will be diluted in a glass of 200 ml soda water added flavour. Placebo consist of 200 ml soda water added the same flavor.
  Bicarbonate/placebo will be prepared in another room by a person not involved in the specific labour. The person will give the drink directly to the woman. Amniotic fluid will be collected and analysed externally.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium bicarbonate (Experimental): Participants receive oral sodium bicarbonate 4.26 gram once.
  Interventions: Drug: Sodium bicarbonate
- Placebo (Placebo Comparator): Participants receive placebo once.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium bicarbonate — 4,26 gram given once.
  Arms: Sodium bicarbonate
Drug: Placebo — Placebo given once.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if oral bicarbonate can treat prolonged labour in nulliparous women with prolonged labour.

The main question it aims to answer is: Do oral bicarbonate and restrictive oxytocin use reduce assisted delivery rate (emergency cesarean and vacuum/forceps delivery) in nulliparous women with prolonged labour.

Researchers will compare bicarbonate and placebo (a look-alike substance that contains no drug) to see if bicarbonate works to treat prolonged labour.

Participants will:

* drink bicarbonate or placebo
* have cervical dilatation reassessed after 2 hours. If still slow progression, they will follow standard protocol for oxytocin augmentation
* will receive a questionnaire 1 month post partum to assess birth experience

1/3 of participants will have amniotic fluid lactate measured at inclusion and after 2 hours

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Danish or English speaking.
* Cephalic presentation.
* Gestational age ≥34+0 - <42+0 (days +weeks) at onset of labour.
* Normal foetal heart rate pattern in the 20 minutes prior to inclusion.
* Spontaneous onset of labour or non-medical induced labour (balloon catheter and/or artificial rupture of membranes).
* Active first stage of labour confirmed, according to Danish national guidelines: Cervical dilatation at ≥4 - <10 cm with regular painful contractions.
* Prolonged labour diagnosed, according to Danish national guidelines: Cervical dilatation progresses at less than 2 cm over a 4-hour period.

Exclusion Criteria:

* Clinical suspicion of infection (2 confirmed temperatures ≥38.5°C with epidural, ≥38 °C without epidural, or broad-spectrum antibiotics initiated)
* Significant medical comorbidity in the form of renal or heart condition, assessed case-by-case basis.
* Serious obstetric complication
* Known allergy or intolerance to sodium bicarbonate.
* Ingestion of sodium bicarbonate in active labour prior to inclusion.
* Current treatment with following medicines: Gabpabpentin, Tetracycline, Ketoconazole (NB! These medications are already generally advised contradicted against induring pregnancy)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 1520 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Difference in incidence of assisted delivery | At birth
  Defined as a composite of emergency caesarean section and instrumental vaginal delivery

SECONDARY OUTCOMES:
Difference in adverse neonatal outcome | From birth until 7 days postpartum
  Composite of perinatal adverse outcomes within the first 7 days of life, including perinatal mortality and neonatal morbidity. Neonatal morbidity is defined as arterial umbilical cord pH <7.10, resuscitation (bag and mask or intubation), hypoxic ischemic encephalopathy II-III, intracranial haemorrhage, neonatal seizures, meconium aspiration syndrome, and admission to a neonatal unit.
Difference in total oxytocin dose | Intrapartum
  Administered intrapartum for augmentation.
Difference in duration of active labour | Intrapartum
  From diagnosis of active labour until childbirth
Difference in birth experience | One month postpartum
  Patient reported using Childbirth Experience Questionnaire (CEQ) which uses a 4-point Likert scale and higher scores indicate a more positive experience.
Difference in amniotic fluid lactate (AFL) concentration | Measured at inclusion and two hours later.
  Collected in the labourroom and analysed externally. Attending clinicians will not know the AFL.
Difference in intra- or postpartum infection | Intrapartum and until 7 days postpartum
  2 confirmed temperatures ≥38.5°C with epidural, ≥38 °C without epidural, or broad-spectrum antibiotics.
Difference in epidural analgesia | Intrapartum
  As documented in the case records
Difference in number of women getting antibiotics during labour | Intrapartum
  As documented in the case records.
Difference in postpartum blood loss | From birth until 24 hours postpartum
  Visual assessment estimated by the attending midwife or calculated using a weight if suspected postpartum haemorrhage.
Difference in women receiving tocolytics used during labour | Intrapartum
  Recorded in the case records
Difference in number of 3rd or 4th-degree perineal tears | Within 2 hours after birth
  Assess by the midwife/doctor suturing the tear.

CONTACTS AND LOCATIONS:
Overall Officials: Nanna Maaløe, PhD, Principal Investigator — University of Copenhagen
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Copenhagen University Hospital, Hvidovre, Copenhagen
  - Copenhagen University Hospital, Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: No